CLINICAL TRIAL: NCT07193927
Title: Investigation of the Efficacy of a Probiotic Mixture in Subjects With Moderate Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): A Mechanistic Trial
Brief Title: Investigation of the Efficacy of a Probiotic Mixture in Moderate Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): A Mechanistic Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AB-MASLD-25
Record Dates: First submitted 2025-08-06; First posted 2025-09-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Fatty Liver Disease, Nonalcoholic; Overweight (BMI > 25)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Lactiplantibacillus plantarum Probiotic Mixture
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo comparator containing maltodextrin

INTERVENTIONS:
Dietary Supplement: Lactiplantibacillus plantarum Probiotic Mixture — A daily oral probiotic capsule containing three specific strains of Lactiplantibacillus plantarum (KABP011, KABP012, KABP013) 1,2 billion CFU with vitamin B1, designed to modulate gut microbiota and improve liver health in MASLD patients. It is compared to a placebo in a 6-month, double-blind, mechanistic trial.
  Arms: Probiotic
Dietary Supplement: Placebo comparator containing maltodextrin — Placebo comparator containing maltodextrin
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate whether a specific probiotic mixture can improve liver health in adults with moderate metabolic dysfunction-associated steatotic liver disease (MASLD).

The main questions it aims to answer are:

Can the probiotics improve liver fat and stiffness as measured by non-invasive imaging (FibroScan® CAP and FAST scores)? Does the probiotic affect other health markers like cholesterol, blood sugar, inflammation, and gut bacteria?

Researchers will compare people taking the probiotic to those taking a placebo (a capsule with no active ingredients) to see if the probiotic has beneficial effects.

Participants will:

Be randomly assigned to take either the probiotic or placebo daily for 6 months.

Attend 3 study visits (at the start, 3 months, and 6 months). Provide blood and stool samples. Undergo liver scans (FibroScan®). Complete a health and nutrition questionnaire.

This study includes adults aged 18-65 with moderate MASLD and certain metabolic health conditions. Participants must not be pregnant, breastfeeding, or taking certain medications or supplements that could interfere with the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 75 years old
* BMI 25 - 38kg/m2
* Diagnosed with MASLD and CAP value > 268 dB/m evaluated by FibroScan®
* High ALT levels (>40 U/L in males and >30 U/L in females)
* Having at least three of the following features compatible with metabolic syndrome:

  i. Waist circumference ≥ 102 cm in males and ≥ 88 cm in females. ii. Fasting serum glucose (≥ 5.6 mmol/L or 100 mg/dl). iii. Glycated haemoglobin (HbA1c ≥ 5.7%/ 39 mmol/L). iv. Diagnosed or treated for type 2 diabetes. v. High blood pressure (≥ 130/85 mmHg). vi. High plasma triglycerides (≥ 1.70 mmol/L or 150 mg/dl). vii. Lower plasma of High-Density Lipoprotein (HDL cholesterol) (≤ 1.0 mmol/L or 40 mg/dl for males and ≤ 1.3 mmol/L or 50 mg/dl for females).
* Stable weight in the last 3 months (less than ± 4% weight variation).
* Stable medication or intake of food supplements for a medical condition that can affect study outcomes according to the Investigator's judgement in the last three months prior to study entry (bile salt sequestrants are not permitted).
* Not planning to change their dietary and lifestyle habits during the study.
* Willing and able to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Fibrosis scores equal or higher than F2 (≥ 8.0 kPa).
* History of acute or chronic hepatitis A, B or C, autoimmune hepatitis, drug-induced liver diseases, severe liver diseases.
* Prior or pending liver transplantation.

Patients with at least one of the following concurrent conditions:

i. Type I diabetes ii. Uncontrolled type II diabetes (HbA1c >8%) iii. Hypertriglyceridemia > 350mg/dl iv. Human Immunodeficiency Virus (HIV) infection v. Diagnosis of hemochromatosis

* Current use of pioglitazone, SGLT-2 inhibitors, or approved drugs for MASLD or steatohepatitis within 8 weeks.
* Current use of bile salt sequestrants within 8 weeks.
* Significant gastrointestinal disease, such as inframmatory bowel disease (IBD, short bowel syndrome, chronic or recurrent diarrhoea, coeliac condition.
* Pancreatic failure, biliary dysfunction (including cholecystectomy and blood bilirubin abnormalities)
* Thyroid dysfunction, as assessed by the investigator (clinical criteria)
* History of:

  i. Cardiovascular disease (ischemic heart disease, heart failure, cerebrovascular disease, periphreal vascular disease).

ii. Cancer or immunosuppression. iii. Gastrointestinal surgery in the previous year (with the exception of appendicitis).

* Patients with a history of chronic alcohol or drug abuse: > 14 units/week for females and > 21 units/week for male
* Chronic and heavy smoking (>20 cigarettes a day)
* Regular intake (> 3 days/week) of other probiotics (including food complements or diary foods with other probiotic strains, e.g. Activia®, Actimel® or similar).
* Intake of nutraceuticals with an effect on hepatic function such as > 500 mg/day omega-3 fatty acids, high-dose vitamin E supplements or milk thistle (sylibum marianum) extract ot their active ingredients (silymarin, silybin) regularly (> 7 days) in the 15 days before study entry.
* Current use of systemic corticosteroids, androgens, clopidogrel, digoxin, acenocoumarol, warfarin, phenytoin, topiramate, lithium, tricyclic antidepressants, MAOIs or second-generation antipsychotics, amiodarone, tamixofen and/or diltiazem.
* History of use (> 3 days) of oral or parenteral antibiotics one month before the study initiation.
* Chronic use of laxatives.
* Debilitating illnesses (advanced liver or kidney disease, severe depression, psychotic symptoms, neurological diseases).
* Current pregnancy (positive urine test) or planning to become pregnant during the study.
* Breastfeeding at the time of eligibility assessment.
* Patients who have participated in a clinical trial in the six-month period before the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in MASLD from baseline | From enrollment to the end of treatment at 6 months.
  Evaluated by CAP (controlled attenuation parameter, dB/m) and FAST score [determined with FibroScan®]

SECONDARY OUTCOMES:
Changes from baseline in Liver Fibrosis (kPa) | From enrollment to the end of treatment at 6 months.
Changes form baseline in MASLD related index - FLI | From enrollment to the end of treatment at 6 months.
  Evaluated by Fatty Liver Index (FLI)
Changes form baseline in MASLD related index - FIB-4 | From enrollment to the end of treatment at 6 months.
  Evaluated by Fibrosis 4 score (FIB-4)
Changes form baseline in MASLD related index - APRI | From enrollment to the end of treatment at 6 months.
  Evaluated by Aspartate aminotransferase-to-platelet ratio index (APRI)
Changes from baseline in metabolic syndrome score (siMS) | From enrollment to the end of treatment at 6 months.
Changes from baseline in weight (kg) | From enrollment to the end of treatment at 6 months.
Changes from baseline in height (cm) | From enrollment to the end of treatment at 6 months.
Changes from baseline in Body Mass Index (BMI) | From enrollment to the end of treatment at 6 months.
  Body Mass Index (BMI) is a person's weight (kg) divided by the square of height (m).
Changes from baseline in waist circumference (cm) | From enrollment to the end of treatment at 6 months.
Changes from baseline in hip circumference (cm) | From enrollment to the end of treatment at 6 months.
Changes from baseline in waist/hip ratio | From enrollment to the end of treatment at 6 months.
  Waist/hip ratio is measured as the waist circumference (cm) divided by the hip circumference (cm).
Changes from baseline in systolic and diastolic blood pressure. | From entollment to the end of treatment at 6 months.
Changes from baseline in serum analysis of blood-based cell profile. | From enrollment to the end of treatment at 6 months.
  Blood count red cell line, white cell line, and platelet line.
Changes from baseline in serum liver enzyme concentrations | From enrollment to the end of treatment at 6 months.
  Aspartate aminotransferase (AST), alanine aminotransferase (ALT), γ-glutamyl transferase (GGT), alkaline phosphatase (AP)
Changes from baseline in serum analysis insulin resistance-related variables | From enrollment to the end of treatment at 6 months.
  Fasting serum glucose, insulin, glycosylated haemoglobin (HbA1c)
Changes from baseline in serum analysis of cholesterol and fatty acid concentrations: | From enrollment to the end of treatment at 6 months.
  Total cholesterol, low-density lipoprotein, high-density lipoprotein, cholesterol, triglycerides.
Changes from baseline in serum analysis of high-sensitivity C-reactive protein (hsCRP) concentration. | From enrollment to the end of treatment at 6 months.
Changes from baseline in serum analysis of albumin concentration | From enrollment to the end of treatment at 6 months.
Changes from baseline in serum analysis of total bilirubin (TBIL) | From enrollment to the end of treatment at 6 months.
Changes from baseline in serum analysis of kidney function biomarkers | From enrollment to the end of treatment at 6 months.
  Uric acid, creatinine (CREA), and blood urea nitrogen (BUN)
Changes from baseline in serum analysis of thyroid hormones | From enrollment to the end of treatment at 6 months.
  Thyrotropin (TSH), thyroxine (T4), triiodothyronine (T3), parathyroid hormone (PTH)
Changes from baseline in serum analysis of iron binding capacity | From enrollment to the end of treatment at 6 months.
  Ferritin, transferrin, binding capacity
Changes from baseline in serum analysis of electrolytes | From enrollment to the end of treatment at 6 months.
  Sodium (Na), potassium (K), chloride (Cl)
Changes from baseline in serum analysis of estimated glomerular filtration rate | From enrollment to the end of treatment at 6 months.
  Estimated glomerular filtration rate (eGFR) measurements developed by the Chronic Kidney Disease Epidemiology (CKD-EPI) collaboration research group.
Changes from baseline in serum analysis of nutritional and metabolic biomarkers | From enrollment to the end of treatment at 6 months.
  Magnesium (Mg), phosphate (P), iron (Fe), calcium (Ca), total protein, cortisol, 25-hydroxyvitamin D.
Changes from baseline in serum metabolite profile by Elevated Global metabolome analysis (amine/phenol and acid channels CIL LC-MS profiling) | From enrollment to the end of treatment at 6 months.
  Quantification of metabolites (around 850 or more), with a minimum confidence of 90% in the identifications.
Changes from baseline in gut microbiota diversity | From enrollment to the end of treatment at 6 months.
  Evaluated through shot gun metagenomics 10GB/spl (Sample QC + Nextera DNA XT (META) Library and NovaSeqX150PE 10 Gb/sample.
Changes from baseline in gut microbiota relative abundance | From enrollment to the end of treatment at 6 months.
  Evaluated through shot gun metagenomics 10GB/spl (Sample QC + Nextera DNA XT (META) Library and NovaSeqX150PE 10 Gb/sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Dr. Josep Trueta, Girona, Girona, Spain